CLINICAL TRIAL: NCT00000856
Title: A Phase I/II Pilot Treatment Study Of CSF Penetration And Response To Ganciclovir And Foscarnet In CMV Neurologic Disease.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 305; 11280 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Encephalopathy; HIV Infections; Radiculitis
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Drug Therapy, Combination; Encephalitis; Foscarnet; Cytomegalovirus Infections; Antiviral Agents; Radiculopathy
MeSH Terms: conditions — Brain Diseases; HIV Infections; Radiculopathy; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Encephalitis; Cytomegalovirus Infections | interventions — Foscarnet; Ganciclovir

INTERVENTIONS:
Drug: Foscarnet sodium
Drug: Ganciclovir

SUMMARY:
To determine the safety and CSF penetration of combined ganciclovir and foscarnet treatment for presumed cytomegalovirus encephalitis or radiculomyelopathy.

This study proposes to investigate the use of combined ganciclovir and foscarnet to maximize the antiviral regimen. Current evidence suggests that a combination of ganciclovir and foscarnet may be the most efficacious therapy and appears to be well tolerated. This study will provide key information regarding safety and CSF penetration of the drugs available for treatment of these lethal diseases. It will also provide preliminary information regarding virologic factors relevant to CMV CNS disease. The study will also provide further data about the natural history of CMV brain infection detected by a combination of symptom complex and PCR identification of CMV in CSF and the potential of semi-quantitative PCR evaluation of the CSF for the disease.

DETAILED DESCRIPTION:
This study proposes to investigate the use of combined ganciclovir and foscarnet to maximize the antiviral regimen. Current evidence suggests that a combination of ganciclovir and foscarnet may be the most efficacious therapy and appears to be well tolerated. This study will provide key information regarding safety and CSF penetration of the drugs available for treatment of these lethal diseases. It will also provide preliminary information regarding virologic factors relevant to CMV CNS disease. The study will also provide further data about the natural history of CMV brain infection detected by a combination of symptom complex and PCR identification of CMV in CSF and the potential of semi-quantitative PCR evaluation of the CSF for the disease.

Patients will be stratified by clinical syndrome as having either primarily A) encephalitis; or B) radiculomyelitis. If patient has combined encephalitis and radiculomyelitis, then the patient will be stratified as encephalitis. CMV therapy with ganciclovir and foscarnet will first be given at an induction level and then a maintenance level. For the first 4 weeks, patients will be given foscarnet plus ganciclovir. Then for the following 20 weeks, patients will be given foscarnet plus ganciclovir with ganciclovir at a lower dose. NOTE: A maximum of 10 patients that have proven to be intolerant to either foscarnet or ganciclovir may receive the alternate agent alone.

NOTE: Ganciclovir experienced subjects will be given GCV at induction and maintenance doses if tolerated.

NOTE: Induction doses will not be re-started in the face of clinical relapse on switching to maintenance therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Patients with treated, stable toxoplasmosis encephalitis with documented stable CT or MR scans may be enrolled if maintenance suppressive therapy is continued.

Patients must have:

* Documented HIV infection.
* Encephalopathy or radiculomyelitis.
* CSF positive for CMV by PCR.
* Signed informed consent from a parent or legal guardian for patients < 18 years.
* CSF cytological analysis should be obtained at the time of enrollment or within 2 weeks prior to enrollment.

NOTE:

* Co-enrollment is encouraged where study procedures do not conflict. Protocols investigating antiviral regimens with potential activity against CMV or other human herpes viruses will be ineligible.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Active CNS infection or malignancy, other than due to CMV or HIV.
* A positive CSF VDRL.
* Any evidence of active disease such as a substantial increase in cryptococcal antigen titer or positive culture. However, patients may be enrolled with stable, treated cryptococcal meningitis.
* A dermatomal or disseminated varicella-zoster infection within 30 days prior to enrollment.
* An active, symptomatic systemic infection, other tan HIV or CMV, for which the patient is not receiving stable therapy for at least 30 days.
* Any other advanced disease likely to cause death in <6 months.
* Known intolerance to both foscarnet and ganciclovir.
* Inability to safely perform a lumbar puncture.

Concurrent Medication:

Excluded:

* Patients on prophylactic antiviral therapy at the time of study enrollment will not be allowed to continue this medication during the study. In the event of the appearance of HSV or VZV infections after enrollment in the study that require systemic therapy, acyclovir or other appropriate medication may be instituted.
* Patients may not receive ZDV therapy during the initial 4 weeks of the study. Concurrent ZDV therapy will be started during maintenance therapy if tolerated. Bone marrow sparing antiretroviral therapy may be used at the investigator's discretion.

NOTE:

* Concurrent medications should be kept to a minimum because of possible interference with the assessment of both safety and pharmacokinetics. But medications absolutely necessary for the subject's welfare may be administered at the discretion of the investigator.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford D, Study Chair; Tselis A, Study Chair

REFERENCES:
- [Background] Smart T. Responding to CMV neurologic infections. GMHC Treat Issues. 1996 Nov;10(11):5-7, 10. PMID 11364010